CLINICAL TRIAL: NCT04361838
Title: Impact of Multi-Denominational Prayer on Morbidity and Mortality of Patients Admitted to the Intensive Care Unite With Corona Virus Infection
Brief Title: The COVID-19 ICU PRAYER Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to the low enrollment, this study is closed. Analysis of data is not performed.
Sponsor: Kansas City Heart Rhythm Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Covid Prayer Study
Record Dates: First submitted 2020-04-16; First posted 2020-04-24 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2021-02

CONDITIONS: Coronavirus Infection
MeSH Terms: conditions — Coronavirus Infections | interventions — Faith Healing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Prayer (Active Comparator): Patients will receive a daily prayer and standard of care treatment from multi-denominational group while in the ICU.
  Interventions: Behavioral: prayer
- No Prayer (No Intervention): Patients will receive standard of care treatment while in the ICU.

INTERVENTIONS:
Behavioral: prayer — receive prayers daily while in ICU
  Arms: Prayer

SUMMARY:
This is a multicenter; double blind randomized controlled study investigating the role of remote intercessory multi-denominational prayer on clinical outcomes in COVID-19 + patients in the intensive care unit. All patients enrolled will be randomized to use of prayer vs. no prayer in a 1:1 ratio. Each patient randomized to the prayer arm will receive a "universal" prayer offered by 5 religious denominations (Christianity, Hinduism, Islam, Judaism and Buddhism) in addition to standard of care. Whereas the patients randomized to the control arm will receive standard of care outlined by their medical teams. During ICU stay, patients will have serial assessment of multi-organ function and APACHE-II/SOFA scores serial evaluation performed on a daily basis until discharge. Data assessed include those listed below.

ELIGIBILITY:
Inclusion Criteria:

* Male or female greater than 18 years of age
* Confirmed positive for COVID-19
* Patient admitted to Intensive Care Unit

Exclusion Criteria:

* Patients admitted to ICU for diagnosis that is not COVID-19 positive.

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-05-21 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Impact of multi-denominational prayer on clinical outcomes of critically ill COVID-19 patients in the Intensive Care Unit on mortality. | daily until patient recovers and moves out of ICU or exits the study, up to 30 days
  This study will measure the difference in mortality of COVID-19 patients who are admitted to ICU - given prayer vs no prayer as an adjunct to standard therapy.

SECONDARY OUTCOMES:
Difference in patient outcomes - Acute Physiology and Chronic Health Enquiry. APACHE II score. | daily until patient recovers and moves out of ICU or exits the study, up to 30 days.
  APACHE II uses 0-71 scale, the higher the score the higher the risk for mortality.
Difference in patient outcomes - Sequential Organ Failure Assessment - SOFA Score | daily until patient recovers and moves out of ICU or exits the study, up to 30 days
  The higher the SOFA score the increased likelihood of organ failure.
Difference in patient outcomes - Length of stay in ICU. | daily until patient recovers and moves out of ICU or exits the study, up to 30 days
  A prolonged length of time in ICU increases mortality.
Difference in patient outcomes - Length of ventilator support | daily until patient recovers and moves out of ICU or exits the study, up to 30 days
  A prolonged length of time with ventilator support increases mortality.
Difference in patient outcomes - length of vasopressor support | daily until patient recovers and moves out of ICU or exits the study, up to 30 days
  A prolonged length of time with vasopressor support increases recovery time.

CONTACTS AND LOCATIONS:
Overall Officials: Dhanunjaya Lakkireddy, MD, Principal Investigator — Kansas City Heart Rhythm Institute
Locations (1):
- Research Medical Center, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koenig HG, Cohen HJ, Blazer DG, Pieper C, Meador KG, Shelp F, Goli V, DiPasquale B. Religious coping and depression among elderly, hospitalized medically ill men. Am J Psychiatry. 1992 Dec;149(12):1693-700. doi: 10.1176/ajp.149.12.1693. PMID 1443246
- [Background] Koenig HG, George LK, Hays JC, Larson DB, Cohen HJ, Blazer DG. The relationship between religious activities and blood pressure in older adults. Int J Psychiatry Med. 1998;28(2):189-213. doi: 10.2190/75JM-J234-5JKN-4DQD. PMID 9724889
- [Background] Currier JM, Foster JD, Witvliet CV, Abernethy AD, Root Luna LM, Schnitker SA, VanHarn K, Carter J. Spiritual struggles and mental health outcomes in a spiritually integrated inpatient program. J Affect Disord. 2019 Apr 15;249:127-135. doi: 10.1016/j.jad.2019.02.012. Epub 2019 Feb 6. PMID 30772739
- [Background] Naimi E, Eilami O, Babuei A, Rezaei K, Moslemirad M. The Effect of Religious Intervention Using Prayer for Quality of Life and Psychological Status of Patients with Permanent Pacemaker. J Relig Health. 2020 Apr;59(2):920-927. doi: 10.1007/s10943-018-0698-8. PMID 30218372
- [Background] Byrd RC. Positive therapeutic effects of intercessory prayer in a coronary care unit population. South Med J. 1988 Jul;81(7):826-9. doi: 10.1097/00007611-198807000-00005. PMID 3393937
- [Background] Harris WS, Gowda M, Kolb JW, Strychacz CP, Vacek JL, Jones PG, Forker A, O'Keefe JH, McCallister BD. A randomized, controlled trial of the effects of remote, intercessory prayer on outcomes in patients admitted to the coronary care unit. Arch Intern Med. 1999 Oct 25;159(19):2273-8. doi: 10.1001/archinte.159.19.2273. PMID 10547166
- [Background] Lakkireddy D, Vacek J, Harris W, Gowda M, Pendyala K, Murray C. Modified Mid America Heart Institute Coronary Care Unit scoring system--a new comprehensive prognostic index for Coronary Care Unit patients. Med Sci Monit. 2005 Mar;11(3):CR95-9. PMID 15735569
- [Background] Jentzer JC, Bennett C, Wiley BM, Murphree DH, Keegan MT, Gajic O, Wright RS, Barsness GW. Predictive Value of the Sequential Organ Failure Assessment Score for Mortality in a Contemporary Cardiac Intensive Care Unit Population. J Am Heart Assoc. 2018 Mar 10;7(6):e008169. doi: 10.1161/JAHA.117.008169. PMID 29525785
- [Background] Yoon JC, Kim YJ, Lee YJ, Ryoo SM, Sohn CH, Seo DW, Lee YS, Lee JH, Lim KS, Kim WY. Serial evaluation of SOFA and APACHE II scores to predict neurologic outcomes of out-of-hospital cardiac arrest survivors with targeted temperature management. PLoS One. 2018 Apr 5;13(4):e0195628. doi: 10.1371/journal.pone.0195628. eCollection 2018. PMID 29621337
- [Background] Yang Y, Peng F, Wang R, Yange M, Guan K, Jiang T, Xu G, Sun J, Chang C. The deadly coronaviruses: The 2003 SARS pandemic and the 2020 novel coronavirus epidemic in China. J Autoimmun. 2020 May;109:102434. doi: 10.1016/j.jaut.2020.102434. Epub 2020 Mar 3. PMID 32143990